CLINICAL TRIAL: NCT04414891
Title: A Randomized Controlled Trial of Non-invasive Ventilation With Adaptive Support Ventilation Versus Neurally Adjusted Ventilator Assist in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Non Invasive Ventilation With NAVA vs ASV for AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAVA_ASV_AECOPD
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Acute Exacerbation of COPD
Keywords: AECOPD; NIV; NAVA; ASV
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Consecutive patients enrolled would be randomized to either the NAVA arm or ASV arm.
  NAVA NIV NAVA will be administered using Servo-i ventilator (Maquet, Getinge Group, Sweden) ASV NIV ASV will be administered using a Galileo GOLD ventilator (Hamilton Medical, AG, Switzerland)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVA arm (Experimental): Delivery of NIV-NAVA NIV NAVA will be administered using Servo-i ventilator (Maquet, Getinge Group, Sweden) with software to compensate for air leaks.
  Subjects randomised to this arm will undergo placement of Edi catheter and will be initiated on NIV. Appropriate NAVA level will be selected based on the scalars corresponding to stable ventilation in pressure support mode. During NAVA, the NAVA level would be increased in multiples of 0.2 cm H2O/µV to attain favourable response (tidal volume 6-8mL/kg RR ≤25). Once the patient's clinical condition stabilises, and the Edi maximum starts declining or remains unchanged with stable tidal volumes, NAVA level will be decreased in steps of 0.2 cm H2O/μV every 2 hours. If response to new settings is not favourable earlier settings will be restored. If favourable response is attained the weaning is continued until peak pressure is <12cm H20 and PEEP requirement is <5cm H2O. NIV will be replaced by a venture mask to titrate SpO2 between 88-92%
  Interventions: Device: Non invasive ventilation
- ASV arm (Active Comparator): Patients randomised to the ASV arm will receive NIV using a Galileo GOLD ventilator (Hamilton Medical, AG, Switzerland). The patients will be ventilated with an initial setting of 100%-minute volume (MV%). Increments of 10% will be made every 15 minutes to achieve clinical response (relief of dyspnea, RR<30, and tidal volume 6-8mL/kg). The expiratory trigger sensitivity will be set at 35% and adjusted accordingly. PEEP will be commenced at 3-4 cm H2O and increased by 1 cm of H2O to achieve SpO2 between 89-92% and maximum PEEP of 10 cm of H2O. Weaning would be performed by reducing the MV% gradually in decrements of 10%/hour to a MV% of 60% after the peak inspiratory pressure decreases to <8 cm of H2O, and the respiratory rate is < 28 breaths per minute and patient is able to maintain SpO2 > 90% at FiO2< 30%. Once the patient is comfortable on these settings, NIV will be replaced with oxygen supplementation using a venturi mask to maintain SpO2 between 89 and 92%.
  Interventions: Device: Non invasive ventilation

INTERVENTIONS:
Device: Non invasive ventilation — Non invasive ventilation will be delivered using an oro-facial interface in both arms. NIV NAVA will be administered using Servo-i ventilator (Maquet, Getinge Group, Sweden) with software to compensate for air leaks.
  ASV arm will receive NIV using a Galileo GOLD ventilator (Hamilton Medical, AG, Switzerland).
  Other Names: NIV

SUMMARY:
Non invasive ventilation is the standard of care in managing patients with exacerbation of chronic obstructive pulmonary disease. However no optimal mode of NIV delivery is established; failure rates remain high, attributed to asynchrony and leak associated with NIV. Neurally adjust ventilator assist is a new mode that may improve patient ventilator interactions, improve synchrony and contribute to improved outcomes. Likewise ASV is a mode principled on the closed loop system and is associated with reduction of work associated with breathing and improved outcomes. In this randomised, non-blinded trial, we study these two modes of NIV delivery in patients of AECOPD with hypothesis being that better synchrony with NAVA may translate to better clinical outcomes.

DETAILED DESCRIPTION:
Study hypothesis We hypothesize that NIV-NAVA would be superior to ASV in reducing the NIV failure rates in patients with AECOPD. In this study, we plan to compare the ASV with NAVA during NIV in patients with AECOPD.

Methods All consecutive patients meeting the inclusion criteria will be screened and assessed for eligibility. Informed consent will be sought and those enrolled would be randomized to to receive NIV using either the ASV or the NIV-NAVA mode. The NIV will be delivered using a oro-nasal mask with supplemental oxygen as needed.

Delivery of NAVA NAVA will be delivered using Servo-i ventilator (Maquet, Getinge Group, Sweden) with software to compensate for air leaks.

NAVA initiation would involve calibration of the Edi module, placement of the nava catheter nasogastrically, verification of position and selecting appropriate nava level on the basis of required pressure support. In case a favourable response is not obtained, NAVA level will beincreased by 0.2 cm/µV until favourable response is seen (tidal volume 6-8mL/kg, respiratory rate < 25/min)

Delivery of ASV ASV will be delivered using a Galileo GOLD ventilator (Hamilton Medical, AG, Switzerland).The patients will be ventilated with an initial setting of 100%-minute volume and will be titrated in increments of 10% as per clinical parameters (respiratory rate, tidal volume).

Monitoring All the patients will be monitored every 15 minutes for respiratory rate, heart rate, blood pressure, Glasgow coma score, pulse oximetry, and signs of respiratory fatigue (paradox), fit of mask and any peri-mask leak. Arterial blood gas analysis will be done at initiation of NIV and then at 1 hour, 4 hours and 24 hours and then at least once a day till primary end point is met.

All the subjects will receive standard of care for acute exacerbation of COPD regardless of their allotted treatment arm.

Randomization Randomization will be done by a computer-generated sequence with blocks of 8 to receive non-invasive ventilation using either the ASV or NAVA. The order of randomisation will be sealed in an opaque envelope, and opened by the physician not directly involved in the study or analysis, at the time of recruitment of patient.

Statistical analysis Results will be presented in a descriptive fashion as mean ± standard deviation (SD), median (interquartile range) or number and percentage. The differences between means of continuous and categorical variables will be analysed using the Student-t-test and chi-square tests, respectively. For data that is not normally distributed the data will be analysed using non-parametric test (Mann-Whitney U).Trends in clinical (respiratory rate and mean arterial blood pressure), arterial blood gas parameters (pH, PaO2, PaCO2) and NIV parameters (peak inspiratory pressure, PEEP, tidal volume) will be analyzed using mixed model technique for repeated measures analysis of variance; the within-groups factor will be time (baseline, one, four and 24 hours), and the between-groups factor will be NIV success. A P value of <0.05 will indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

Consecutive subjects with AECOPD will be eligible for inclusion in the study if they meet all the following: (a) an acute (<7 days) sustained worsening of any of the patient's respiratory symptoms (cough, sputum quantity or character, dyspnea) beyond the normal day-to-day variation; (b) arterial blood gas analysis showing a PaCO2 >45 mm Hg with either pH between 7.10 and 7.35 or respiratory rate (fR) >30 breaths/minute; and, (c) exclusion of other causes of acute breathlessness such as acute heart failure, pulmonary embolism, pneumonia, and pneumothorax.

Exclusion Criteria:

Patients with any one of the following criteria will be excluded from the current study:

1. Non-COPD acute hyper-capneic respiratory failure
2. Hypotension (systolic blood pressure <90 mmHg)
3. Severe impairment of consciousness (Glasgow coma scale score <8)
4. Inability to clear respiratory secretions
5. Abnormalities that preclude proper fit of the NIV interface (agitated or uncooperative patient, facial trauma or burns, facial surgery, or facial anatomical abnormality
6. Subjects who have an artificial airway like tracheostomy tube or T-tube
7. Contraindications for insertion of naso-/orogastric feeding tube (facial/nasal trauma, recent upper airway surgery, esophageal surgery, esophageal varices, upper gastrointestinal bleeding)
8. Unwillingness to undergo placement of nasogastric catheter
9. Known phrenic nerve lesions
10. Suspected diaphragmatic weakness
11. Patient already on home NIV therapy for chronic respiratory failure
12. Failure to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of NIV failure | From initiation of NIV to either intubation or re-initiation of NIV or successful weaning
  NIV failure will be considered in case of
  • Endotracheal intubation

SECONDARY OUTCOMES:
28-day mortality rate | 28 days
  28-day mortality including ICU and hospital deaths will be assessed
90-day mortality rate | 90 days
  90-day mortality including deaths after discharge
Time to NIV failure | 28 days
  From initiation of NIV to either intubation or re-initiation of NIV
Time to successful weaning | 28 days
  Time to successful weaning will be defined as the duration between initiation of NIV and successful weaning from NIV
Physician's ease of use of the mode on visual analogue scale | Assessed every 8 hours until primary outcome
  Ease of use will be recorded on a scale of 100 mm, with 0 being very easy and 100 very difficult
Patient assessed level of comfort using visual analogue scale | 28 days
  Level of comfort will be assessed on a scale of 100 mm, 0 being very comfortable and 100 very uncomfortable
Average number of manipulations | 28 days
  Assessed daily for 5 days or until primary outcome whichever occurs first
Asynchrony index | 28 days
  Assessed daily until primary outcome or 5 day period, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Inderpaul Singh Sehgal, MD DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Respiratory Intensive Care Unit, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sehgal IS, Kalpakam H, Dhooria S, Aggarwal AN, Prasad KT, Agarwal R. A Randomized Controlled Trial of Noninvasive Ventilation with Pressure Support Ventilation and Adaptive Support Ventilation in Acute Exacerbation of COPD: A Feasibility Study. COPD. 2019 Apr;16(2):168-173. doi: 10.1080/15412555.2019.1620716. Epub 2019 Jun 4. PMID 31161812
- [Background] Chen C, Wen T, Liao W. Neurally adjusted ventilatory assist versus pressure support ventilation in patient-ventilator interaction and clinical outcomes: a meta-analysis of clinical trials. Ann Transl Med. 2019 Aug;7(16):382. doi: 10.21037/atm.2019.07.60. PMID 31555696
- [Background] Tajamul S, Hadda V, Madan K, Tiwari P, Mittal S, Khan MA, Mohan A, Guleria R. Neurally-Adjusted Ventilatory Assist Versus Noninvasive Pressure Support Ventilation in COPD Exacerbation: The NAVA-NICE Trial. Respir Care. 2020 Jan;65(1):53-61. doi: 10.4187/respcare.07122. Epub 2019 Oct 22. PMID 31641071
- [Background] Sehgal IS, Dhooria S, Aggarwal AN, Behera D, Agarwal R. Asynchrony index in pressure support ventilation (PSV) versus neurally adjusted ventilator assist (NAVA) during non-invasive ventilation (NIV) for respiratory failure: systematic review and meta-analysis. Intensive Care Med. 2016 Nov;42(11):1813-1815. doi: 10.1007/s00134-016-4508-z. Epub 2016 Aug 25. No abstract available. PMID 27562243
- [Background] Wang DQ, Luo J, Xiong XH, Zhu LH, Zhang WW. [Effect of non-invasive NAVA on the patients with acute exacerbation of chronic obstructive pulmonary disease]. Zhonghua Yi Xue Za Zhi. 2016 Nov 15;96(42):3375-3378. doi: 10.3760/cma.j.issn.0376-2491.2016.42.004. Chinese. PMID 27866528
- [Derived] Chhabria BA, Prasad KT, Dhooria S, Muthu V, Aggarwal AN, Agarwal R, Gandra RR, Sehgal IS. A randomized controlled trial comparing non-invasive ventilation delivered using neurally adjusted ventilator assist (NAVA) or adaptive support ventilation (ASV) in patients with acute exacerbation of chronic obstructive pulmonary disease. J Crit Care. 2023 Jun;75:154250. doi: 10.1016/j.jcrc.2022.154250. Epub 2023 Jan 19. PMID 36680884